CLINICAL TRIAL: NCT05861531
Title: The Combined Association of an Oral Motor Stimulation and Language Intervention on Preterm Infant Feeding
Brief Title: Combined Oral Motor Stimulation and Language on Preterm Infant Feeding
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Julia Mayne, Assistant Professor of Pediatrics, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2015266
Record Dates: First submitted 2023-04-24; First posted 2023-05-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-07

CONDITIONS: Language Delay; Language Development; Feeding; Difficult, Newborn; Mother-Infant Interaction; Maternal Behavior
Keywords: Neonatal feeding; Neonatal language; Oromotor stimulation; Newborn reading; Parent infant interaction; LENA
MeSH Terms: conditions — Language Development Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Statistician will analyze deidentified data and Bayley assessments will be conducted by blinded psychologists.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oral motor stimulation with language (Experimental): 1. Obtain baseline LENA recording 2. Review language curriculum and provide LENA linguistic feedback 3. LENA recording every 2 weeks until 36 weeks corrected 4. Review age-appropriate language curriculum and provide LENA linguistic feedback from prior weeks 5. When reaches 33-34 weeks postmenstrual age and medically stable, occupational therapists will conduct 10-15 minute oral motor stimulation prior to a feeding time for 10 total days over a 2 week period 6. Final LENA feedback and PTSD screen
  Assessments: 1. PSS:NICU at 36 weeks corrected 2. PPQ screen at 7, 12, and 24 months corrected 3. Child Behavior Checklist at 24 months corrected 4. Bayley Scales of Infant and Toddler Development at 12 and 24 months
  Interventions: Behavioral: Oromotor stimulation; Behavioral: Reading curriculum; Behavioral: LENA recording; Behavioral: LENA linguistic feedback
- Oral motor stimulation (Active Comparator): 1. Obtain baseline LENA recording 2. LENA recording every 2 weeks until 36 weeks corrected 3. When reaches 33-34 weeks postmenstrual age and medically stable, occupational therapists will conduct 10-15 minute oral motor stimulation prior to a feeding time for 10 total days over a 2 week period. 4. Final LENA feedback and PTSD screen.
  Assessments: 1. PSS:NICU at 36 weeks corrected 2. PPQ screen at 7, 12, and 24 months corrected 3. Child Behavior Checklist at 24 months corrected 4. Bayley Scales of Infant and Toddler Development at 12 and 24 months
  Interventions: Behavioral: Reading curriculum; Behavioral: LENA recording; Behavioral: LENA linguistic feedback; Behavioral: No oromotor stimulation
- Standard Care (No Intervention): 1. Obtain baseline LENA recording 2. LENA recording every 2 weeks until 36 weeks corrected 3. 6. Final LENA feedback and PTSD screen
  Assessments: 1. PSS:NICU at 36 weeks corrected 2. PPQ screen at 7, 12, and 24 months corrected 3. Child Behavior Checklist at 24 months corrected 4. Bayley Scales of Infant and Toddler Development at 12 and 24 months

INTERVENTIONS:
Behavioral: Oromotor stimulation — This will begin around 33 weeks corrected, the day following the first NTrainer measurements. The oral stimulation program will be modeled after the protocol designed and studied for preterm infants and will be implemented for a goal of 10 consecutive days within a 14 day period. This includes 10 minutes of stroking the cheeks, lips, gums, and tongue, and the final 5 minutes consisting of mid tongue stroking, eliciting a suck with gloved finger, and sucking on a pacifier provided in the NICU. This will occur 15-30 minutes before a scheduled tube feeding when the infant is tolerating bolus enteral feeds of 120 ml/kg/day for at least 48 hours. This will occur behind a curtain to ensure blinding of staff and parents. Modifications will be made for infants that remain intubated and only 10 minutes of the stroking of the cheeks, lips, gums, and tongue will occur. Stimulation will cease if episodes of oxygen desaturation and/or apnea/bradycardia occur during the stimulation.
  Arms: Oral motor stimulation with language
Behavioral: Reading curriculum — Written packets with biweekly lessons. The first two lessons include how to begin to read and talk to their baby. The second two lessons include reading or talking about the day using infant directed speech. The final two lessons include continuing to engage with the baby through interactive reading.
  Arms: Oral motor stimulation; Oral motor stimulation with language
Behavioral: LENA recording — The LENA device provides 24 hours of language recordings placed inside an infant vest. The recordings are uploaded to a computer which analyzes total adult word counts, infant vocalizations, conversational turns, background noise, and silence.
  Arms: Oral motor stimulation; Oral motor stimulation with language
Behavioral: LENA linguistic feedback — LENA recordings of adult word counts, infant vocalizations, and conversational turns will be provided in printed form after each recording with review of each recording and progress over time.
  Arms: Oral motor stimulation; Oral motor stimulation with language
Behavioral: No oromotor stimulation — This will begin around 33 weeks corrected, the day following the first NTrainer measurements. The standard care group will not receive any stimulation but will have a study personnel present behind a curtain to ensure blinding of family, staff, and investigators. The study personnel will remain behind a curtain for 10-15 minutes prior to a feed for 10 days over a 14-day period beginning when the infant is tolerated 120 mL/kg/day for at least 48 hours.
  Arms: Oral motor stimulation

SUMMARY:
This is a randomized controlled trial to study an oromotor stimulation in combination with a reading curriculum in the NICU among preterm infants using oral muscle exercises, Language Environment Analysis (LENA) recordings, linguistic feedback, and a language curriculum to improve the neonatal inpatient oral feeding and language outcomes for preterm infants.

DETAILED DESCRIPTION:
This project aims to determine the effects of an oral motor stimulation combined with a reading curriculum vs an oral motor stimulation alone vs controls among preterm infants born 23-30 weeks gestation in the NICU. We hypothesize that the infants receiving an oral motor stimulation in conjunction with a reading curriculum will start oral feeding at an earlier age, have fewer days to full oral feeding, and fewer days in the NICU compared to infants receiving an oral motor stimulation and controls. We hypothesize that the infants receiving an oral motor stimulation in conjunction with a reading curriculum will have increased infant vocalizations, increased conversational turns, increased adult word counts, decreased maternal stress, decreased degree of post-traumatic stress post-discharge, improved receptive and expressive language development at 12 and 24 months, and improved parent reported behavioral outcomes at 24 months.

ELIGIBILITY:
Inclusion Criteria:

* 23-30 weeks
* English and Spanish speaking

Exclusion Criteria:

* Major congenital anomalies
* Surgical necrotizing enterocolitis
* Non-English and Non-Spanish speaking

Ages: 23 Weeks to 30 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 124 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
Oral feeding measures | From date of birth to day of NICU hospital discharge
  Days to first oral feeding, days to complete oral feeding, hospital days

SECONDARY OUTCOMES:
Number of adult, infant, and conversational turn word counts measured by LENA device | From enrollment and biweekly until 36 weeks corrected
  Adult word counts, conversational turns, and infant vocalizations from each recording
Maternal stress | 36 weeks corrected
  Using the Parental Stressor Scale: Neonatal Intensive Care Unit (PSS:NICU) to understand the parents' perceptions of stress within the NICU using 46 questions on a Likert scale with a 5 as extremely stressful and 1 as not stressful at all. Not applicable is also an option as well.
Maternal post traumatic stress disorder | 7, 12 and 24 months
  Perinatal posttraumatic stress disorder (PTSD) Questionnaire to measure maternal PTSD. PTSD symptoms of subjects will be measured with the modified PPQ, which consists of 14 items that measure three dimensions: unwanted intrusions or re-experiencing of delivery, avoidance or emotional numbing and hyperarousal. In the modified PPQ, each PPQ item is rated on five-point Likert scale (with a score of 0 indicating not sick to 4 indicating very sick). mothers with modified PPQ scores⩾19 and <19 as having and not having PTSD, respectively.
Child Behavior | 24 months
  Using Child Behavior Checklist to measure child behavioral and emotional problems in childhood
Bayley Scales of Infant and Toddler Development, Fourth Edition | 12 months and 24 months
  Individual assessment used to assess development of infants between 1 to 42 months of age. Domains are as follows: cognitive, language, motor, social-emotional, and adaptive behavior. Scores can be used to assess infants progress over time. Mean scores of 100 with 1 standard deviation below the mean indicating mild delay and 2 standard deivations below the mean indicating moderate to severe delay.

CONTACTS AND LOCATIONS:
Locations (1):
- Women & Infants NICU, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fucile S, Gisel EG, McFarland DH, Lau C. Oral and non-oral sensorimotor interventions enhance oral feeding performance in preterm infants. Dev Med Child Neurol. 2011 Sep;53(9):829-835. doi: 10.1111/j.1469-8749.2011.04023.x. Epub 2011 Jun 27. PMID 21707601
- [Background] Adams-Chapman I, Bann CM, Vaucher YE, Stoll BJ; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Association between feeding difficulties and language delay in preterm infants using Bayley Scales of Infant Development-Third Edition. J Pediatr. 2013 Sep;163(3):680-5.e1-3. doi: 10.1016/j.jpeds.2013.03.006. Epub 2013 Apr 10. PMID 23582139
- [Background] Dudek-Shriber L. Parent stress in the neonatal intensive care unit and the influence of parent and infant characteristics. Am J Occup Ther. 2004 Sep-Oct;58(5):509-20. doi: 10.5014/ajot.58.5.509. PMID 15481778
- [Background] Callahan JL, Borja SE, Hynan MT. Modification of the Perinatal PTSD Questionnaire to enhance clinical utility. J Perinatol. 2006 Sep;26(9):533-9. doi: 10.1038/sj.jp.7211562. Epub 2006 Jul 6. PMID 16826190